CLINICAL TRIAL: NCT01310686
Title: Genotypic Evaluation of Chronic Exudative Macular Degeneration Despite Monthly Anti-Vascular Endothelial Growth Factor (VEGF) Therapy
Brief Title: Genetics Study of Wet Age-Related Macular Degeneration (AMD) Non-Responders to Vascular Endothelial Growth Factor (VEGF) Therapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: West Coast Retina Medical Group, Inc. (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Arthur D. Fu, MD, Principal Investigator, West Coast Retina Medical Group, Inc.
Other Study IDs: FVF4990s
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Wet AMD
Keywords: wet AMD anti-VEGF; Genetic analysis of patients with Wet AMD who have not responded fully to anti-VEGF treatments

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Wet AMD Non-Responders to Anti-VEGF

SUMMARY:
To obtain a genotypic analysis of patients with chronic exudative age-related macular degeneration noted to have subretinal or intraretinal edema despite continuous monthly Anti-VEGF therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent for participation in this study
* Subjects diagnoses of neovascular AMD who are on a monthly anti-VEGF regimen (have had >10 or more ranibizumab and/or bevacizumab injections within the last year) and who still have intra-retinal or subretinal fluid as confirmed by the Investigator

Exclusion Criteria:

* Subjects with a Pigment Epithelial Detachment Exclusively
* Subjects with Serous Pigment Epithelial Detachments
* Subjects with history of the following:

idiopathic polypoidal choroidal vasculopathy

* pathologic degenerative myopia
* central serous chorioretinopathy
* familial drusen
* adult onset foveal pattern dystrophy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Wet Age-Related Macular Degeneration
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-04; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Genetic analysis of patients with chronic wet age-related macular degeneration despite continuous anti-VEGF treatment | This is a one time only blood draw.

SECONDARY OUTCOMES:
To evaluate demographic and clinical characteristics in patients treated with anti-VEGF therapy who fail to respond completely. | This is a one time only blood draw and assessment of clinical characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- West Coast Retina Medical Group, Inc., San Francisco, California, United States